CLINICAL TRIAL: NCT02405585
Title: An Exploratory Phase 2 Study of Neoadjuvant Chemotherapy Followed by Stereotactic Body Radiation Therapy (SBRT) With Algenpantucel-L (HyperAcute®-Pancreas) Immunotherapy in Subjects With Borderline Resectable Pancreatic Cancer
Brief Title: Immunotherapy and SBRT Study in Borderline Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0605; 1409-1350 (Other: Office of Biotechnology Activities)
Record Dates: First submitted 2015-03-25; First posted 2015-04-01 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer; Pancreatic Carcinoma Non-resectable
Keywords: Pancreatic Cancer; Immunotherapy; Vaccine Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mFOLFIRINOX + Algenpantucel-L (HAPa) Immunotherapy (Experimental): SOC mFOLFIRINOX + Algenpantucel-L (HAPa) Immunotherapy
  Day 93-100 Disease evaluated: Progressive disease = salvage therapy off study. Day 93-100 Disease evaluated: Stable disease or better = SBRT + HAPa on days 1 and 15 of radiotherapy Post SBRT: surgery + adjuvant SOC Gemcitabine + HAPa given 1 and 15 for 6 cycles.
  Post adjuvant therapy: 6 monthly immunizations with HAPa
  Interventions: Drug: mFOLFIRINOX; Biological: Algenpantucel-L Immunotherapy; Radiation: SBRT; Drug: Gemcitabine

INTERVENTIONS:
Drug: mFOLFIRINOX — mFOLFIRINOX consisting of Oxaliplatin 85 mg/m^2 IV over 2 hours; Irinotecan 180 mg/m^2 IV over 90 minutes; Leucovorin 400 mg/m^2 IV over 2 hours; Fluorouracil 2.4 g/m^2 IV over 46 hours - given on days 15, 29, 43, 57, 71 and 85
  Other Names: Oxaliplatin; Eloxatin®; Irinotecan; Camptosar®; Leucovorin; Citrovorum factor; folinic acid; Fluorouracil; 5-Fluorouracil; 5-FU
Biological: Algenpantucel-L Immunotherapy — HAPa1 and HAPa2 immunotherapy components Algenpantucel-L Immunotherapy (HAPa) consisting of 300 Million HAPa cells given by intradermal injection for up to 28 doses total.
  Other Names: HyperAcute®-Pancreas; HAPa
Radiation: SBRT — Subjects that have at least stable disease at evaluation (day 93-100) are eligible to receive SBRT radiation given at 1.8 Gy per fraction for 28 fractions for a total dose of 50.4 Gy.
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 given intravenously over 30 minutes for 3 weeks (days 1, 8 and 15) with 1 week rest.
  Given as adjuvant treatment (days 1, 8 and 15) with 1 week rest for 6 cycles after surgical resection.
  Other Names: Gemzar

SUMMARY:
Unfortunately, despite the best clinical efforts and breakthroughs in biotechnology, most patients diagnosed with pancreatic cancer continue to die from the rapid progression of their disease. One primary reason for this is that the disease is typically without symptoms until significant local and/or distant spread has occurred and is often beyond the chance for cure at the time of the diagnosis. The lack of any treatment to substantially increase long term survival rates is reflected by the poor outcomes associated with this disease, specifically time to disease progression and overall survival.

However, another important part of the body is now being looked at as a target for therapy against this disease - the immune system. Scientists have clearly shown that pancreatic tumor cells produce a number of defective proteins, or express normal proteins in highly uncharacteristic ways, as part of this cancer. In some cancers, these abnormalities can cause an immune response to the cancer cells much in the way one responds to infected tissue. In progressive cancers however, the immune system fails to effectively identify or respond to these abnormalities and the cancer cells are not attacked or destroyed for reasons not yet fully understood. This clinical trial proposes a new way to stimulate the immune system to recognize pancreatic cancer cells and to stimulate an immune response that destroys or blocks the growth of the cancer.

This new method of treatment helps the immune system of pancreatic cancer patients to "identify" the cancerous tissue so that it can be eliminated from the body. As an example, patients with certain diseases may require an organ transplant to replace a damaged kidney or heart. After receiving their transplant, these patients receive special drugs because they are at great danger of having an immune response that destroys or "rejects" the transplanted organ. This "rejection" occurs when their immune system responds to differences between the cells of the transplanted organ and their own immune system by attacking the foreign tissue in the same way as it would attack infected tissue. When the differences between foreign tissues and the patient's body are even larger, as with the differences between organs from different species, the rejection is very rapid, highly destructive, and the immunity it generates is longlasting. This is called hyperacute rejection and the medicine used to immunize patients in this protocol tries to harness this response to teach a patient's immune system to fight their pancreatic cancer just as the body would learn to reject a transplanted organ from an animal.

To do this, Algenpantucel-L immunotherapy contains human pancreatic cancer cells that contain a mouse gene that marks the cancer cells as foreign to patient's immune systems. The immune system therefore attacks these cancer cells just as they would attack any truly foreign tissue, destroying as much as it can. Additionally, the immune system is stimulated to identify differences (aside from the mouse gene) between these cancer cells and normal human tissue as foreign. This "education" of the immune system helps treat the patient because pancreatic cancer cells already present in a treated patient are believed to show some of the same differences from normal tissue as the modified pancreatic cancer cells in the product. Due to these similarities, the immune system, once "educated" by the Algenpantucel-L immunotherapy, identifies the patient's cancer as foreign and attacks.

Historically, external beam radiation has been part of the treatment of pancreatic cancer, both before and after surgical resection. Recent breakthroughs in technology now allow for more intensive doses of radiation to be delivered to the body with greater precision. These newer, more precise radiation treatments, called stereotactic body radiation, deliver more intensive radiation to a locally advanced tumor and are now being employed in the treatment of pancreatic cancer. Stereotactic body radiation may increase the chances that surgery will successfully remove a pancreatic cancer.

In this experimental study, all patients will be given a strong combination of antitumor chemotherapy while receiving injections of an immunotherapy drug consisting of two types of pancreatic cancer cells that have been modified to make them more easily recognized and attacked by the immune system. The investigators propose to test this new treatment paradigm along with stereotactic body radiation in patients with borderline resectable pancreatic cancer to demonstrate that treatment with this combination of therapies increases the time until the tumor progresses as well as overall survival.

DETAILED DESCRIPTION:
This protocol attempts to treat pancreatic cancer using a naturally occurring barrier to xenotransplantation in humans to increase the efficacy of immunizing subjects against their pancreatic cancer. In this protocol, the transfer of the murine alpha(1,3)galactosyltransferase [alpha(1,3)GT] gene to immunotherapy component cells results in the cell surface expression of alpha(1,3)galactosyl-epitopes (alpha gal) epitopes on membrane glycoproteins and glycolipids. These epitopes are the major target of the hyperacute rejection response. This response occurs when organs are transplanted from lower animal donor species into primates and results in rapid destruction of transplanted tissue and an augmented response against transplant antigens, including antigens not related to the alpha gal epitopes. Human hosts have pre-existing anti-alpha-gal antibodies that are thought to result from chronic immunological stimulation due to exposure to alpha-gal epitopes that are naturally expressed on normal gut flora and these antibodies may comprise up to 1% of serum IgG. Opsonization and lysis of the immunotherapy component cells mediated by this antibody is believed to increase the efficiency of antigen processing by targeting vaccine components to antigen presenting cells via the Fc gamma receptor.

ELIGIBILITY:
Inclusion Criteria:

* A histological diagnosis of adenocarcinoma of the pancreas confirmed by pathology.
* Patients must have borderline resectable pancreatic cancer with no metastatic spread as determined by a baseline diagnostic CT scan with intravenous contrast (or MRI). CT should be performed according to a defined pancreas protocol such as triphasic cross-sectional imaging with thin slices. Optimal multi-phase technique including a non-contrast phase plus arterial, pancreatic parenchymal and portal venous phase of contrast enhancement with thin cuts (3mm) throughout the abdomen is preferred. Studies must be evaluated by a radiologist and/or surgeon and deemed borderline resectable as defined below:

  1. Borderline resectable- Tumors considered borderline resectable are defined as follows:
  2. Venous involvement of the SMV/portal vein demonstrating tumor abutment with impingement and narrowing of the lumen, encasement of the SMV/portal vein but without encasement of the nearby arteries, or short-segment venous occlusion resulting from either tumor thrombus or encasement but with suitable vessel proximal and distal to the area of vessel involvement, allowing for safe resection and reconstruction
  3. Gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery without extension to the celiac axis.
  4. Tumor abutment of the SMA not to exceed greater than 180 degrees of the circumference of the vessel wall.
* Tumors considered to be unresectable due to local advancement include an absence of distant metastases as well as:

  1. Head: Greater than 180 degrees SMA encasement or any celiac abutment or unreconstructible SMV/portal occlusion or aortic invasion or encasement.
  2. Body: Greater than 180 degrees SMA or celiac encasement or unreconstructible SMV/portal occlusion or aortic invasion.
  3. Tail: SMA or celiac encasement greater than 180 degrees.
  4. Nodal status: Involvement of lymph nodes beyond the field of resection should be considered unresectable due to distant spread and therefore not eligible for this protocol.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Serum albumin ≥ 2.0 gm/dL.
* Expected survival ≥ 6 months.
* Adequate organ function including:

  1. Marrow: WBC ≥3000/mm^3 and platelets ≥100,000/mm^3.
  2. Hepatic: serum total bilirubin ≤ 1.5 mg/dL, ALT (SGPT) and AST (SGOT) ≤3 x upper limit of normal (ULN) at time of enrollment. If a patient has elevated liver function tests at the time of initial presentation or develops them during work-up and they are the result of a mechanical obstruction of biliary drainage by tumor compression or invasion, a biliary drain may be placed as described in NCCN Practice Guidelines in Oncology V2.2012. If drainage allows for the liver function tests to come within inclusion criteria, the patient may be enrolled.
  3. Renal: serum creatinine (sCr) ≤2.0 x ULN, or creatinine clearance (Ccr) ≥30 mL/min.
* Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* All subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product, and for one month after the last immunization.

Exclusion Criteria:

* Age <18-years-old.
* Active metastases.
* Other malignancy within five years, unless the probability of recurrence of the prior malignancy is <5% as determined by the Principal Investigator based on available information. Patient's curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant.
* Current, active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subjects taking chronic systemic corticosteroid therapy for any reason are not eligible. Subjects may receive steroids as prophylactic anti-emetics per the mFOLFIRINOX regimen. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require chronic systemic corticosteroids after beginning treatment, will be removed from study.
* Significant or uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias within the last six months.
* Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Autoimmune disease (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), etc.). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., active liver cirrhosis) or a serious illness in medical opinion of the clinical investigator.
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.).
* A known history of allergy or hypersensitivity to any of the study drugs or any of their excipients.
* Pregnant or nursing women due to the unknown effects of immunization on the developing fetus or newborn infant. (For patients with child bearing potential, a βHCG must be completed within 14 days of first treatment).
* Known HIV positive.
* Prior treatment with chemotherapy or radiation for pancreatic cancer or prior treatment with radiation for other diagnoses to expected pancreatic cancer treatment fields.
* Current grade II or higher peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 18 months (assuming enrollment period of 1 year)
  The primary objective of this study is to assess progression free survival after treatment with a regimen of mFOLFIRINOX with algenpantucel-L immunotherapy followed by SBRT in subjects who have borderline resectable pancreatic cancer.

SECONDARY OUTCOMES:
Overall Survival | 30 months (assuming enrollment period of 1 year)
  A secondary objective of this study is to assess overall survival (OS) in pancreatic cancer patients with borderline resectable pancreatic cancer who will receive a regimen of mFOLFIRINOX with algenpantucel-L Immunotherapy followed by SBRT.
Frequency and grade of adverse events of FOLFIRINOX in combination with algenpantucel-L Immunotherapy | 18 months (assuming enrollment period of 1 year)
  A secondary objective of this study is to assess the safety (frequency and grade of adverse events) of administration of algenpantucel-L Immunotherapy given in combination with a standard of care regimen of chemotherapy mFOLFIRINOX followed by SBRT
Immune Response | 18 months (assuming enrollment period of 1 year)
  A secondary objective of this study is to assess the immunologic responses of subjects with pancreatic cancer undergoing antitumor immunization with algenpantucel-L Immunotherapy as measured by anti-alpha Gal antibodies, and-tumor antibodies, and total IgE.
Tumor Response | 18 months (assuming enrollment period of 1 year)
  A secondary objective of this study is to assess the tumor response rate as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and Immune Response Criteria (irRC).
Resection Rate | 18 months (assuming enrollment period of 1 year)
  A secondary objective of this study is to assess the R0 resection rate following neoadjuvant chemotherapy, immunotherapy and SBRT.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Louisville, Louisville, Kentucky
  - Lahey Clinic, Burlington, Massachusetts
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Seattle Cancer Care Alliance, Seattle, Washington